CLINICAL TRIAL: NCT04375748
Title: Hospital Registry of Acute Myocarditis: Evolution of the Proportion of Positive SARS-COV-2 Cases During the Covid-19 Pandemic, Case Characteristics and Prognoses
Brief Title: Hospital Registry of Acute Myocarditis: Evolution of the Proportion of Positive SARS-COV-2 (COVID19) Cases
Acronym: MYOCOVID
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0139
Record Dates: First submitted 2020-04-21; First posted 2020-05-05 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Acute Myocarditis
Keywords: Covid19; Myocarditis; Epidemiology; Prognosis; Mortality
MeSH Terms: conditions — COVID-19; Myocarditis | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated for symptoms of acute myocarditis.: Patients treated in intensive coronary care unit (ICCU) or intensive care unit (ICU), in one of the participating hospitals, for symptoms of acute myocarditis confirmed by a myocardial MRI and/or a CT scan and/or a myocardial biopsy.
  Interventions: Diagnostic Test: Performing routine care (clinical and paraclinical tests); Diagnostic Test: Examinations for the research:

INTERVENTIONS:
Diagnostic Test: Performing routine care (clinical and paraclinical tests) — ECG, standard biology and cardiology tests, and routine transthoracic echocardiography (TTE), MRI
Diagnostic Test: Examinations for the research: — Systematic research by polymerase chain reaction (PCR) for Covid-19 in the blood and in an oro-pharyngeal swab, in addition to the usual immunologic, bacteriological, viral and parasitic tests carried out as part of the routine care of all patients with suspected myocarditis.
  A 30-days phone call follow-up (vital status) and a systematic 1-year follow-up will be realized (clinic, biology, ECG, TTE, +/- MRI)

SUMMARY:
To date, the effects of SARS-Cov-2 (Covid-19) on the myocardium and the role it plays in the evolution towards an acute myocarditis are badly understood. The current pandemic of this emerging virus is an opportunity to assess the proportion of acute myocarditis attributable to SARS-Cov-2(Covid-19) and to assess the clinical, biological and imaging presentations, by means of a national prospective multicentre hospital registry of cases of acute myocarditis.

DETAILED DESCRIPTION:
Although research on the subject has only recently started developing, the links have already been described between SARS-Cov-2 infection, the severity of the clinical status, and the presence of risk factors or a history of cardiovascular disease (hypertension, diabetes, stroke, etc.). Additionally, depending on the series and definition used for cardiac injury (troponin elevation and/or natriuretic peptides), this concerns 7-29% of patients with a clear predominance in severe patients. The mechanisms behind these troponin elevations and cardiac injury are likely to be multiple and variable depending on clinical presentation,severity and patient history. A significant association was found between troponin elevation, and that of CRP and NtproBNP, suggesting an inflammatory part to this cardiac damage. As with other coronaviruses, SARS-Cov-2 infection can cause massive release of proinflammatory cytokines which can lead to inflammation of the vascular wall. This can be the cause of true instability or even rupture of plaque(type1 infarction) but can also be responsible for tissue hypoxia without rupture of plaque causing myocardial pain (infarction type 2). In addition, there may be areal myocardial inflammation causing acute myocarditis, secondary to the cytokine storm or direct damage to the myocardium by the virus itself. In case of acute coronary syndrome presentation, a coronary exploration should be realized to highlight or eliminate a type 1 infarction, but it is clearly difficult to distinguish between a type 2 suffering (no viral attack direct but suffering from hypotension or hypoxia for example) and inflammatory myocardial damage with or without direct viral myocardial damage (myocarditis). In the context of the viral pandemic at Covid19, although few data exist,it is legitimate to consider the possibility of true arrays of acute inflammatory myocarditis or by direct viral attack which could thus modify the natural history and the prognosis of patients, thus justifying a dedicated diagnosis and treatment. The primary objective was to assess the proportion of positive SARS-Cov-2 cases among the patients included (hospitalized for acute myocarditis). During the study period, this proportion will be assessed at regular intervals, for example every month, or more frequently if the number of patients included varies substantially from one week to another. This will make it possible to trace a development curve for the entire period of the pandemic.

The secondary objectives were (1) to describe the clinical, biological and imaging characteristics of the acute myocarditis among the positive and negative SARS-Cov-2 patients of the myocarditis cohort; (2) to assess the short-term (30 days) and long-term (1 year) prognosis of the acute myocarditis among the positive and negative SARS-Cov-2 patients of the myocarditis cohort and (3) to identify the factors associated with a 30-day and 1-year prognosis of cases of acute myocarditis.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated in ICCU or ICU (polyvalent, surgical or medical), in one of the participating hospitals, for symptoms of acute myocarditis confirmed by a myocardial MRI and/or a CT scan and/or a myocardial biopsy. It seems important to include elderly patients who may be under guardianship or curatorship since these patients seem to present the most severe forms. Additionally, the populations most affected by viral myocarditis are generally adolescents and young adults,which justifies including them in the study too. Pregnant women are a population at potentially greater risk, particularly during the third trimester because of the neuro-hormonal changes inherent in pregnancy. This justifies trying to implement the investigator's knowledge through this observational study.

Exclusion Criteria:

* Refusal to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated in ICCU or ICU (polyvalent, surgical or medical), in one of the participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 756 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Evolution of the proportion of positive SARS-COV-2 cases. | 6 months.
  Estimate at hospital discharge, over a period of 6 months, the evolution of the proportion of positive SARS-COV-2 cases among patients hospitalized for acute myocarditis in Intensive Cardiac Care Unit or Intensive Care Unit (polyvalent, surgical or medical), in the 19 hospitals participating in the study.

SECONDARY OUTCOMES:
Ultrasound characteristics. | 1 year
  Describe at the admission and during the treatment ultrasound characteristics of the acute myocarditis among the positive and negative SARS-Cov-2 patients of the myocarditis cohort; Echocardiographic parameters: Volumes (mm3)
Ultrasound characteristics. | 1 year
  Describe at the admission and during the treatment ultrasound characteristics of the acute myocarditis among the positive and negative SARS-Cov-2 patients of the myocarditis cohort ; Echocardiographic parameters: diameters (mm)
Ultrasound characteristics. | 1 year
  Describe at the admission and during the treatment ultrasound characteristics of the acute myocarditis among the positive and negative SARS-Cov-2 patients of the myocarditis cohort (Echocardiographic parameters: ventricular diastolic function (mm);
Ultrasound characteristics. | 1 year
  Describe at the admission and during the treatment ultrasound characteristics of the acute myocarditis among the positive and negative SARS-Cov-2 patients of the myocarditis cohort (Echocardiographic parameters: ventricular systolic function (mm);
Ultrasound characteristics. | 1 year
  Describe at the admission and during the treatment ultrasound characteristics of the acute myocarditis among the positive and negative SARS-Cov-2 patients of the myocarditis cohort ; Echocardiographic parameters: Left atrium volume (mm3);
Ultrasound characteristics. | 1 year
  Describe at the admission and during the treatment ultrasound characteristics of the acute myocarditis among the positive and negative SARS-Cov-2 patients of the myocarditis cohort ; Echocardiographic parameters: Maximum velocity of tricuspid valve insufficiency;
Ultrasound characteristics. | 1 year
  Describe at the admission and during the treatment ultrasound characteristics of the acute myocarditis among the positive and negative SARS-Cov-2 patients of the myocarditis cohort ; Echocardiographic parameters: Presence and quantification of a valvular regurgitation
Ultrasound characteristics. | 1 year
  Describe at the admission and during the treatment ultrasound characteristics of the acute myocarditis among the positive and negative SARS-Cov-2 patients of the myocarditis cohort ; Echocardiographic parameters: Presence of a pericardial effusion
Assess prognosis of the acute myocarditis . | The short-term (30 days) and long-term (1 year).
  Assess the short-term (30 days) and long-term (1 year) prognosis of the acute myocarditis among the positive and negative SARS-Cov-2 patients of the myocarditis cohort. The 30-day prognosis will be defined in function to the outcome: A death, whatever the cause, A cardiovascular arrest with recovery, A cardiogenic shock, An acute lung oedema or One of the events cited above.
  The 1-year prognosis will be defined in function to the outcome: A death, whatever the cause, The need to resort to transplantation and/or chronic assistance, A rehospitalization for cardiovascular reasons (heart failure, painful relapse, recovered cardiac arrest, myocarditis relapse, ACS), A myocarditis relapse, or one of the events cited above. The 1-year prognosis will also be defined in function to the New York Heart Association
  (NYHA) class.
The factors associated with acute myocarditis cases . | The short-term (30 days) and long-term (1 year).
  Identify the factors associated with a 30-day and 1-year prognosis of cases of acute myocarditis cardiovascular (Terminal heart failure, Acute edema of the lung, Cardiogenic shock, Sudden death / Ventricular rhythm disorder Pulmonary embolism, Aortic dissection Infectious endocarditis Stroke) or no cardiovascular (Acute respiratory syndrome, septic shock of non-cardiac origin, cancer, Public road accident, end-stage respiratory failure, insufficiency, end-stage renal Failure)
Biological characteristics | 1 year
  Describe the biological parameters on admission and during the treatment (troponinemia (ng/ml)
Biological characteristics | 1 year
  Describe the biological parameters on admission and during the treatment NtproBNP(pg/ml)
Biological characteristics | 1 year
  Describe the biological parameters on admission and during the treatment CRP(mg/ml)
Describe at the admission and during the treatment cardiac MRI parameters | 1 year
  Ventricular volumes (ml)
Describe at the admission and during the treatment cardiac MRI parameters | 1 year
  Systole Diameter
Describe at the admission and during the treatment cardiac MRI parameters | 1 year
  Diastole Diameter
Describe at the admission and during the treatment cardiac MRI parameters | 1 year
  Longitudinal deformation of left ventricle;
Describe at the admission and during the treatment cardiac MRI parameters | 1 year
  Longitudinal deformation of right ventricle;
Describe at the admission and during the treatment cardiac MRI parameters | 1 year
  Total volume of left ventricular oedema
Describe at the admission and during the treatment cardiac MRI parameters | 1 year
  Quantification of T2 before contrast agent
Describe at the admission and during the treatment cardiac MRI parameters | 1 year
  Quantification of T1 before contrast agent
Describe at the admission and during the treatment cardiac MRI parameters | 1 year
  Perfusion anomalies
Describe at the admission and during the treatment cardiac MRI parameters | 1 year
  Total volume of early left ventricular alteration
Describe at the admission and during the treatment cardiac MRI parameters | 1 year
  Total volume of late left ventricular alteration
Describe at the admission and during the treatment cardiac MRI parameters | 1 year
  Quantification of T1 after contrast agent
Describe at the admission and during the treatment cardiac MRI parameters | 1 year
  Presence of a pericardial effusion

CONTACTS AND LOCATIONS:
Overall Officials: Clément Delmas, Principal Investigator — CHU Toulouse, Hôpital Rangueil
Locations (65):
- France (62):
  - Cardiology, Aix-en-Provence
  - Reanimation, Amiens
  - Cardiology, Angers
  - Reanimation, Angers
  - Cardiology, Avignon
  - Cardiology, Bordeaux
  - Pediatric cardiology, Bordeaux
  - Reanimation, Bordeaux
  - Cardiology, Brest
  - Cardiology, Caen
  - Pediatric Cardiology, Caen
  - Cardiology, Clermont-Ferrand
  - Pediatric cardilogy, Clermont-Ferrand
  - Reanimation, Clermont-Ferrand
  - Pediatric cardiology, Dijon
  - Cardiology, Grenoble
  - Pediatric cardiology, Grenoble
  - Reanimation, Grenoble
  - Cardiology, Lille
  - Pediatric cardiology, Lille
  - Pediatric cardiology, Limoges
  - Cardiology, Lyon
  - Pediatric cardiology, Lyon
  - Cardiology, Marseille
  - Pediatric cardiology, Marseille
  - Cardiology, Metz
  - Cardiology, Montpellier
  - Millénaire Clinical - Cardiology, Montpellier
  - Pediatric cardiology, Montpellier
  - Reanimation, Montpellier
  - Cardiology, Nancy
  - Pediatric cardiology, Nancy
  - Cardiology, Nantes
  - Pediatric cardiology, Nantes
  - Cardiology, Nice
  - Pediatric cardiology, Nice
  - Cardiology, Nîmes
  - Cardiology, Henri Mondor Hospital, Paris
  - Cardiology, Paris
  - Henri Mondor Hospital Reanimation, Paris
  - Marie Lannelongue Hospital - Pediatric Cardiology, Paris
  - Marie Lannelongue Hospital Cardiology, Paris
  - Reanimation, Paris
  - Robert Debré Hospital - Pediatric cardiology, Paris
  - Saint Antoine Hospital - Cardiology, Paris
  - Cardiology, Poitiers
  - Reanimation, Poitiers
  - Pediatric cardiology, Reims
  - Cardiology, Rennes
  - Pediatric reanimation, Rennes
  - Cardiology, Rouen
  - Pediatric cardiology, Rouen
  - Pédiatric cardiology, Strasbourg
  - Reanimation, Strasbourg
  - CHU de TOULOUSE, Toulouse
  - Croix du Sud Clinical, Toulouse
  - Pasteur Clinical - Cardiology, Toulouse
  - Pasteur Clinical - Pediatric cardiology, Toulouse
  - Pediatric Cardiology, Toulouse
  - Cardiolgy, Tours
  - Pediatric Cardiology, Tours
  - Cardiology, Valenciennes
- Cardiology, Martinique, Martinique
- Cardiology, Mamoudzou, Mayotte
- Pédiatric cardiology, Réunion, Reunion